CLINICAL TRIAL: NCT04717518
Title: Anchoring Patients Pain Scores in the Emergency Department
Status: Completed | Type: Observational
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Landry Dorsett, DO, Principal Investigator, CHRISTUS Health
Other Study IDs: 2020-132
Record Dates: First submitted 2020-11-18; First posted 2021-01-22 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Pain; Chest Pain; Headache; Joint Pain; Muscle Pain; Back Pain; Neck Pain
Keywords: Emergency Room
MeSH Terms: conditions — Abdominal Pain; Chest Pain; Headache; Arthralgia; Myalgia; Back Pain; Neck Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Anchor Survey: Patients will likely rate their pain lower.
  Interventions: Other: Measurement of Pain
- Higher Anchor Survey: Patients will likely rate their pain higher.
  Interventions: Other: Measurement of Pain

INTERVENTIONS:
Other: Measurement of Pain — Patients will fill out a brief survey concerning the current visit to the ED.

SUMMARY:
The proposed research will be a prospective, observational study to test the hypothesis that anchoring will affect verbal pain scores in the emergency department. There will be a small retrospective aspect to this study to obtain patient satisfaction ratings.

DETAILED DESCRIPTION:
The investigators will evaluate a convenience sample of patients presenting to the ED with a complaint of pain. Patients will be consented for participation and will fill out a brief survey concerning the current visit in the ED. There will be two forms of the survey. Participants will be randomly assigned to one of the two survey forms. Participants will first be asked if their pain score for this visit is greater than or less than an anchor number provided. In this survey, the investigators will use 20 and 80 as our anchoring numbers. The participants will then have a follow up question asking them to estimate their pain score on a 0-100 scale. Investigators will then perform a chart review to determine patient satisfaction scores for that specific visit to determine if the anchoring effect has any input on patient satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Presenting to the ED with a chief complaint of any type of pain

Exclusion Criteria:

* Under 18 years of age
* Refusal to consent
* Incarcerated patients
* Pregnant patients
* Unable to complete survey secondary to clinical instability, severe pain, or disorientation determined by a study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects include patients presenting to the Emergency Department at CHRISTUS Spohn Shoreline with a chief complaint of pain.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Utilization of a questionnaire to measure the mean pain scores between two intervention groups based on the numeric pain score scale | Through study completion, an average of 1 year
  A questionnaire will be used to measure pain scores by utilizing a numeric pain scale (0-100) and measure the effect of anchoring bias on pain scores in the Emergency Department. It is hypothesized that a lower pain score anchor will lead to a lower reported pain score by the patient.

SECONDARY OUTCOMES:
An analysis to examine the influence of anchoring on patient satisfaction for patients with common chief complaints related to pain in the Emergency Department. It is unknown if anchoring affects a patient's overall satisfaction. | Through study completion, an average of 1 year
  Patients receive Press-Ganey questionnaire to evaluate their visit to the Emergency Department. We will measure if the anchoring pain score affects the patients overall satisfaction with their Emergency Department care.

CONTACTS AND LOCATIONS:
Overall Officials: Landry Dorsett, DO, Principal Investigator — CHRISTUS Spohn Health System
Locations (1):
- CHRISTUS Spohn Health System, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Plans to collaborate with other universities in other studies and/or grants.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] "CDC Guideline for Prescribing Opioids for Chronic Pain." CDC, 2019, www.cdc.gov/drugoverdose/prescribing/guideline.html.
- [Background] Colorado Opioid Safety Pilot Results Report The Colorado Opioid Safety Collaborative Background. Colorado Hospital Association, 2017.
- [Background] "Nonopioid Pain Management | AHA." American Hospital Association, 2018, www.aha.org/bibliographylink-page/2018-09-28-nonopioid-pain-management. Accessed 13 Nov. 2019.
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] "Overdose Death Maps." CDC, 13 Aug. 2019, www.cdc.gov/drugoverdose/data/prescribing/overdosedeath-maps.html.
- [Background] Compton WM, Jones CM, Baldwin GT. Relationship between Nonmedical Prescription-Opioid Use and Heroin Use. N Engl J Med. 2016 Jan 14;374(2):154-63. doi: 10.1056/NEJMra1508490. No abstract available. PMID 26760086
- [Background] Meisel ZF, Lupulescu-Mann N, Charlesworth CJ, Kim H, Sun BC. Conversion to Persistent or High-Risk Opioid Use After a New Prescription From the Emergency Department: Evidence From Washington Medicaid Beneficiaries. Ann Emerg Med. 2019 Nov;74(5):611-621. doi: 10.1016/j.annemergmed.2019.04.007. Epub 2019 Jun 20. PMID 31229392
- [Background] Marco CA, Kanitz W, Jolly M. Pain scores among emergency department (ED) patients: comparison by ED diagnosis. J Emerg Med. 2013 Jan;44(1):46-52. doi: 10.1016/j.jemermed.2012.05.002. Epub 2012 Jul 13. PMID 22795472
- [Background] Marco CA, Nagel J, Klink E, Baehren D. Factors associated with self-reported pain scores among ED patients. Am J Emerg Med. 2012 Feb;30(2):331-7. doi: 10.1016/j.ajem.2010.12.015. Epub 2011 Mar 1. PMID 21367555
- [Background] Tversky A, Kahneman D. Judgment under Uncertainty: Heuristics and Biases. Science. 1974 Sep 27;185(4157):1124-31. doi: 10.1126/science.185.4157.1124. PMID 17835457
- [Background] Northcraft, Gregory B, and Margaret A Neale. "Experts, Amateurs, and Real Estate: An Anchoring-andAdjustment Perspective on Property Pricing Decisions." Organizational Behavior and Human Decision Processes, vol. 39, no. 1, 1987, pp. 84-97, 10.1016/0749-5978(87)90046-x.
- [Background] . Wansink, Brian, et al. "An Anchoring and Adjustment Model of Purchase Quantity Decisions." Journal of Marketing Research, vol. 35, no. 1, Feb. 1998, pp. 71-81, 10.1177/002224379803500108.
- [Background] Yadav, Manjit S. "How Buyers Evaluate Product Bundles: A Model of Anchoring and Adjustment." Journal of Consumer Research, vol. 21, no. 2, Sept. 1994, p. 342, 10.1086/209402.
- [Background] Liang, Hanchao, et al. "Bounded Rationality, Anchoring-and-Adjustment Sentiment, and Asset Pricing." The North American Journal of Economics and Finance, vol. 40, Apr. 2017, pp. 85-102, 10.1016/j.najef.2017.02.001. Accessed 13 Nov. 2019.
- [Background] Brewer NT, Chapman GB, Schwartz JA, Bergus GR. The influence of irrelevant anchors on the judgments and choices of doctors and patients. Med Decis Making. 2007 Mar-Apr;27(2):203-11. doi: 10.1177/0272989X06298595. PMID 17409369
- [Background] Amir R, Leiba R, Eisenberg E. Anchoring the Numeric Pain Scale Changes Pain Intensity Reports in Patients With Chronic But Not With Acute Pain. Pain Pract. 2019 Mar;19(3):283-288. doi: 10.1111/papr.12738. Epub 2018 Nov 20. PMID 30328678
- [Background] Riva P, Rusconi P, Montali L, Cherubini P. The influence of anchoring on pain judgment. J Pain Symptom Manage. 2011 Aug;42(2):265-77. doi: 10.1016/j.jpainsymman.2010.10.264. Epub 2011 Mar 12. PMID 21402456
- [Background] Marco CA, Marco AP, Plewa MC, Buderer N, Bowles J, Lee J. The verbal numeric pain scale: effects of patient education on self-reports of pain. Acad Emerg Med. 2006 Aug;13(8):853-9. doi: 10.1197/j.aem.2006.04.020. PMID 16880501